CLINICAL TRIAL: NCT03319004
Title: Validation of Phase Lag Entropy(PLE) as an Indicator of Depth of Sedation in Patients Undergoing Spinal Anesthesia: Comparative Analysis With Bispectral Index
Brief Title: Validation of Phase Lag Entropy(PLE) as an Indicator of Depth of Sedation in Patients Undergoing Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Dong Woo Han, Principal Investigator, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3-2017-0145
Record Dates: First submitted 2017-10-01; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Surgery Requiring Spinal Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compare bispectral index and phase lag entropy (Experimental)
  Interventions: Device: apply phase lag entropy sensor

INTERVENTIONS:
Device: apply phase lag entropy sensor — apply phase lag entropy sensor as well as bispectral index sensor on forehead during the sedation using propofol

SUMMARY:
For verifying the phase lag entropy as the tool for measurement of level of consciousness, the investigators compared phase lag entropy to bispectral index. Using Target-Controlled Infusion pump, propofol was infused for sedation during the spinal anesthesia. The investigators measured Observer's Assessment of Alertness/Sedation Scale as the propofol concentration rises. At the same time, The investigators observed phase lag entropy score and bispectral index score.

ELIGIBILITY:
Inclusion Criteria:

* patients who require sedation during the spinal anesthesia

Exclusion Criteria:

* dementia, CVA patients, patients have problems with communication

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2017-07-19 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-07-18 (Estimated)

PRIMARY OUTCOMES:
phase lag entropy score | through study completion, an average of 1 year
  phase lag entropy score

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea